CLINICAL TRIAL: NCT00811239
Title: A Controlled Clinical Trial on The Use of a Specific Antivenom Against Envenoming by Bungarus Multicinctus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Collaborators: Karolinska Institutet (Other); Swedish International Development Cooperation Agency (SIDA) (Other Government)
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: antivenom; second study on snakebite
Record Dates: First submitted 2008-12-16; First posted 2008-12-18 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Snake Bite
Keywords: antivenom; snake bite; Bungarus multicinctus; Vietnam
MeSH Terms: conditions — Snake Bites | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (Other): As the antivenom was not yet clinically available until 2006, all patients included during the first two years (2004-2005) received supportive therapy only.
  Interventions: Other: Supportive Care
- antivenom group (Active Comparator): The patients included during the third year (2006) were treated with antivenom therapy and supportive care.
  Interventions: Drug: Bungarus multicinctus-candidus Antivenom

INTERVENTIONS:
Drug: Bungarus multicinctus-candidus Antivenom — Five to ten ampoules of antivenom, depending on severity of muscle paralysis, were diluted with isotonic glucose solution to have total 50 ml and infused intravenously by electric pump during one hour. After a period of 6-8 hours, a second infusion was administered, under similar condition to the first, if no clinical improvement or adverse reaction had been noted. The patients also received supportive care such as intubation, ventilation...if necessary.
  Arms: antivenom group
Other: Supportive Care — Supportive Care only (endotracheal intubation, mechanical ventilation...)
  Arms: control group

SUMMARY:
In northern Vietnam, a vast majority of the most severe envenomed patients are bitten by Bungarus multicinctus. Hitherto, these victims have received supportive care only. The aims of this study were to assess the possible efficacy and side effects of a newly produced antivenom.

DETAILED DESCRIPTION:
Venomous snakebites constitute a serious health problem in many Asian countries. In Vietnam, the burden of snakebite on the public health stimulated Calmette to conduct original studies at the Vaccine Institute in Saigon over a hundred years ago and to develop the first snake antivenom ever.

In northern Vietnam, a vast majority of the most severe envenomed patients are bitten by Bungarus multicinctus, which is the only krait species giving rise to significant morbidity and mortality in the area. Its venom contains toxins which can cause severe neuromuscular blockade but which do not give rise to swelling or necrosis at the site of the bite.

Supportive care is an important part of the management of snakebites, but antivenom administration is the mainstay therapy in the majority of medically significant envenomings. Such specific therapy may dramatically reduce the consequences of the envenomation. In Vietnam, no specific antivenom against B. multicinctus has been available until recently when it has produced for clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Envenomed by B. multicinctus
* Showed clinical signs of systemic envenomation (neuromuscular signs)
* Provided written informed consent (during the year 2006)

Exclusion Criteria:

* Pregnancy
* Patients had a known history of intolerance to equine serum

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2004-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
duration of mechanical ventilation | the length of ICU stay

SECONDARY OUTCOMES:
clinical course during ICU stay | the length of ICU stay
complications (Ventilator associated pneumonia...) | the length of ICU stay
adverse effects (anaphylaxis, serum sickness...) | the length of ICU stay
hyponatremia, renal and liver function | the length of ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Höjer, MD, PhD, Study Director — Karorinska Institute, Swedish Poisons Information Centre
Locations (1):
- Vietnam Poison Control Center, Bach Mai Hospital, HMU, Hanoi, Vietnam

REFERENCES:
- [Result] Chan JC, Cockram CS, Buckley T, Young K, Kay R, Tomlinson B. Evenoming by Bungarus multicinctus (many-banded krait) in Hong Kong. J Trop Med Hyg. 1995 Dec;98(6):457-60. PMID 8544231
- [Result] Pe T, Myint T, Htut A, Htut T, Myint AA, Aung NN. Envenoming by Chinese krait (Bungarus multicinctus) and banded krait (B. fasciatus) in Myanmar. Trans R Soc Trop Med Hyg. 1997 Nov-Dec;91(6):686-8. doi: 10.1016/s0035-9203(97)90524-1. PMID 9509180
- [Result] Cheng AC, Winkel KD. Snakebite and antivenoms in the Asia-Pacific: wokabaut wantaim, raka hebou ("walking together"). Med J Aust. 2001 Dec 3-17;175(11-12):648-51. doi: 10.5694/j.1326-5377.2001.tb143762.x. No abstract available. PMID 11837876
- [Result] Dart RC, McNally J. Efficacy, safety, and use of snake antivenoms in the United States. Ann Emerg Med. 2001 Feb;37(2):181-8. doi: 10.1067/mem.2001.113372. PMID 11174237
- [Result] White J. Envenoming and antivenom use in Australia. Toxicon. 1998 Nov;36(11):1483-92. doi: 10.1016/s0041-0101(98)00138-x. PMID 9792162
- [Result] Karlson-Stiber C, Persson H, Heath A, Smith D, al-Abdulla IH, Sjostrom L. First clinical experiences with specific sheep Fab fragments in snake bite. Report of a multicentre study of Vipera berus envenoming. J Intern Med. 1997 Jan;241(1):53-8. doi: 10.1046/j.1365-2796.1997.80896000.x. PMID 9042094
- [Derived] Ha TH, Hojer J, Trinh XK, Nguyen TD. A controlled clinical trial of a novel antivenom in patients envenomed by Bungarus multicinctus. J Med Toxicol. 2010 Dec;6(4):393-7. doi: 10.1007/s13181-010-0051-4. PMID 20358414